CLINICAL TRIAL: NCT03320187
Title: NITROGLYCERINE SKIN PATCH VS PLACEBO PATCH FOR ENHANCING CERVICAL RIPENING IN LABOR INDUCTION: A RANDOMIZED CONTROLLED TRIAL
Brief Title: Nitroglycerin Skin Patches for Facilitating Cervical Ripening: A Randomized Controlled Trial
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Collaborators: Dr. Ahmed S. Abd El-Hameed (Unknown); Prof. Abdel-Megeeed I. Abdel- Megeeed (Unknown)
Responsible Party: Principal Investigator, Peter Nagy Aziz Hanna, Resident Physician, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OG MS27042017
Record Dates: First submitted 2017-09-22; First posted 2017-10-25 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Induction of Labor Affected Fetus / Newborn
MeSH Terms: interventions — Nitroglycerin; Dinoprostone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group A (Experimental): Nitroglycerin as Nitroderm TTSⓇ skin patch is applied on the upper chest alongside with regular induction of labor protocol ( 3gm/ 8 hours DinoprostoneⓇ vaginal tablet in the posterior vaginal fornix)
  Interventions: Drug: Nitroderm TTS; Drug: Dinoprostone
- Group B (Placebo Comparator): Placebo patch is applied on the upper chest alongside with regular induction of labour protocol ( 3gm/ 8 hours DinoprostoneⓇ vaginal tablet in the posterior vaginal fornix)
  Interventions: Drug: Dinoprostone

INTERVENTIONS:
Drug: Nitroderm TTS — Transdermal nitroglycerin 5mg skin patch
  Other Names: Nitroglycerin transdermal patch
  Arms: Group A
Drug: Dinoprostone — Dinoprostone 3gm vaginal tablet will be used as the study method of labor induction
  Other Names: Prostaglandin E2 Analogue

SUMMARY:
This study aims to establish the efficacy of transdermal glyceryl trinitrate as a nitric oxide donor in addition to dinoprostone for induction of cervical ripening in the third trimester through progression in the Bishop's score during 24 hour period.

DETAILED DESCRIPTION:
Objectives: The primary outcome of the study is to compare the changes occurring to the cervix through the progression in the Bishop's score between NO donor (nitroglycerine patch) vs placebo; in combination with a well-established method of induction (Dinoprostone).

The secondary objective of the study is to observe and report possible fetal and maternal side effects that may be associated. This will establish the safety and tolerability of NO donors.

Research Question: Does the usage of Nitroglycerine skin patch enhance cervical ripening and facilitate induction of labor by Dinoprostone?

Null hypothesis: Nitroglycerine skin patch does not cause advantage for ripening of the cervix nor facilitate the process of labor induction.

Alternative hypothesis : Nitroglycerine skin patch has favorable effect in enhancing cervical ripening and the outcome of induction of labor.

ELIGIBILITY:
Inclusion Criteria:

1. Singleton living full-term fetus.
2. Cephalic presentation,
3. Bishop score less than 5,
4. Assuring fetal monitoring,
5. The mother does not have PROM,

Exclusion Criteria:

1. Expected fetal anomaly (eg. by ultrasound),
2. Abnormal presentation,
3. Multiple pregnancy,
4. Non assuring fetal CTG,
5. Fetus more than 90th percentile of expected weight,
6. Previous maternal obstructed labor or previous cesarean section,
7. Maternal obstetric or medical complication,
8. Structural anomaly of the uterus

Ages: 17 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2016-12; Primary Completion 2017-09 (Actual); Study Completion 2017-09-21 (Actual)

PRIMARY OUTCOMES:
Changes in the cervical Bishop's score | 6,12,18 and 24 hours after administration
  progression of Bishop's score recorded twice during the induction of labor

SECONDARY OUTCOMES:
Development of any fetal or maternal side effects | From the time of administration of medication, cases will be assessed every 6 hours till 24 hours after delivery at time of discharge
  associated headache and nausea (for instance) are well-recognized side effects during the induction of labor
Need of Oxytocin to initiate uterine contractions | from time of patch administration up to 24 hours
  Whether the case managed to initiate uterine contractions without the need to induce them with oxytocin

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Abdel-Megeeed I. Abdel-Megeeed, Doctorate, Study Chair — Ain Shams University Maternity Hospital; Ahmed S. Abd El-Hamid, Doctorate, Study Director — Ain Shams University Maternity Hospital
Locations (1):
- AinShams University Maternity Hospital, Cairo, Egypt

REFERENCES:
- [Result] Sharma Y, Kumar S, Mittal S, Misra R, Dadhwal V. Evaluation of glyceryl trinitrate, misoprostol, and prostaglandin E2 gel for preinduction cervical ripening in term pregnancy. J Obstet Gynaecol Res. 2005 Jun;31(3):210-5. doi: 10.1111/j.1447-0756.2005.00271.x. PMID 15916656
- [Result] Nunes FP, Campos AP, Pedroso SR, Leite CF, Avillez TP, Rodrigues RD, Meirinho M. Intravaginal glyceryl trinitrate and dinoprostone for cervical ripening and induction of labor. Am J Obstet Gynecol. 2006 Apr;194(4):1022-6. doi: 10.1016/j.ajog.2005.10.814. PMID 16580291
- [Result] West HM, Jozwiak M, Dodd JM. Methods of term labour induction for women with a previous caesarean section. Cochrane Database Syst Rev. 2017 Jun 9;6(6):CD009792. doi: 10.1002/14651858.CD009792.pub3. PMID 28599068
- [Result] Kelly AJ, Munson C, Minden L. Nitric oxide donors for cervical ripening and induction of labour. Cochrane Database Syst Rev. 2011 Jun 15;(6):CD006901. doi: 10.1002/14651858.CD006901.pub2. PMID 21678363

DOCUMENTS (2):
  • Study Protocol (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03320187/Prot_000.pdf
  • Informed Consent Form (2017-04-27): https://cdn.clinicaltrials.gov/large-docs/87/NCT03320187/ICF_001.pdf